CLINICAL TRIAL: NCT05057780
Title: Measuring the Impact of an Interactive Communication Skills Curriculum on Internal Medicine Residents: A Cluster Randomized Educational Study
Brief Title: Measuring the Impact of an Interactive Communication Skills Curriculum on Internal Medicine Residents
Acronym: IMCOMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17-1454
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Resident Communication Skills Rated by Patients

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: Resident participants did not know which curriculum was intervention and which was control. Patient participants did not know what communication curriculum their resident physician had completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Curriculum (Experimental): The intervention course consisted of 3 hour-long sessions on communication delivered over a 4-month period. It differed from the control course in subject matter and pedagogy. Subject matter focused on specific skills used in communication: reflective listening, responding to emotion, and providing information within a broad range of communication scenarios. In terms of pedagogy, the intervention course was interactive with a focus on skills practice, communication drills, and improvisation to engage learners. The sessions consisted of fifteen minutes of lecture and 45 minutes of skills practice.
  Interventions: Other: Communication Skills Curriculum
- Control (Standard) Curriculum (Active Comparator): The control course consisted of three hour-long didactic lectures on delivering bad news, discussing prognosis, and talking to patients about pain. The majority of time in these lectures was spent on didactic material. Little, if any, time was spent practicing skills or on interactive skill building. The three parts of the course were delivered over a 4-month period.
  Interventions: Other: Communication Skills Curriculum

INTERVENTIONS:
Other: Communication Skills Curriculum — Our novel intervention adapted curricula around effective skills used to navigate common communication challenges in clinical practice. These skills were selected after determining patterns from multiple communication sessions delivered to over 6,000 healthcare providers. Our main goal was to enhance communication with patients by helping residents gain confidence and competence using these under-utilized communication skills, regardless of the communication challenge. Over the course of three, 1-hour long sessions on communication in the 2017-2018 academic year, internal medicine residents learned three of these highly effective and often under-utilized skills; reflective listening, responding to emotion and reframing, respectively.

SUMMARY:
This study seeks to assess whether a novel method of teaching communication skills is effective in improving the communication skills of internal medicine residents. Effective communication is widely accepted as an essential skill in both clinical practice and post-graduate training. While the body of research on effective communication is maturing, training that incorporates this new data lags behind. Methodological difficulties inherent to the study of communication training programs further complicates the effort to create effective, evidence-based training programs for the next generation of practitioners. Cleveland Clinic has taught its internally developed relationship-centered communication model, the R.E.D.E. Model, to over 7000 providers in less than 5 years. While teaching this course, common communication themes emerged as areas where providers often "get stuck". This proposal details a cluster randomized educational study of a novel communication training curriculum that addresses 3 of the common communication themes that emerged and how those themes occur in multiple, different communication challenges. The curriculum will be delivered to 2nd and 3rd year internal medicine residents over three, 1-hr long training sessions. The investigators' primary aim is to test whether residents trained to identify and communicate through these themes will receive better scores on communication from patients seen in their general internal medicine clinic. The investigators will also assess the effect of this training on patient compliance and on management of common chronic diseases such as hypertension, depression, and diabetes. Lastly, the investigators will measure the effect of the training course on resident self-perceived burnout and empathy.

DETAILED DESCRIPTION:
This trial employed a cluster-randomized design. The residency program randomly divides the residents into 5 groups when they arrive as interns. These groups receive lectures together for all three years of residency and have similar schedules. The investigators used this predetermined structure to randomize the residents' communication course for this study. Two of the five groups were selected using a random number generator to receive the control course and three of the five groups received the intervention course. Although participation in the research study was voluntary, attending the assigned communication course was a mandatory educational activity for the residents.

Control (standard) Course:

The control course consisted of three hour-long didactic lectures on delivering bad news, discussing prognosis, and talking to patients about pain. The majority of time in these lectures was spent on didactic material. Little, if any, time was spent practicing skills or on interactive skill building. The three parts of the course were delivered over a 4-month period.

Intervention Course:

The intervention course also consisted of three hour-long sessions on communication delivered over a 4-month period. It differed from the control course in subject matter and pedagogy. Subject matter focused on specific skills used in communication: reflective listening, responding to emotion, and providing information within a broad range of communication scenarios. In terms of pedagogy, the intervention course was interactive with a focus on skills practice, communication drills, and improvisation to engage learners. The sessions consisted of fifteen minutes of lecture and 45 minutes of skills practice.

Faculty, senior residents, and fellows at the Center for Excellence in Healthcare Communication (CEHC) facilitated the control and intervention courses.33 Instructors at the CEHC taught facilitators best practices in adult learning theory, small and large group facilitation, and effective communication skills. Two trained facilitators led each course. The same facilitators taught the control and intervention courses.

PARTICIPANTS

Resident Participants:

Residents were recruited from Cleveland Clinic's Internal Medicine Residency program from November 2017 through April 2018. A total of 120 residents were eligible to participate in the study as they were post-graduate (PGY) 2 and 3 residents scheduled to receive mandatory educational curriculum on communication. Residents were invited to participate in the study first by an e-mail and again in person immediately prior to the start of the course. Residents received an information sheet about the study which explained that both the residents and their patients would be surveyed. Residents who completed the baseline surveys were considered enrolled, and their patients were sampled as detailed below. Residents were given a $10 gift card in compensation for their time and effort. While participation in the study was optional, all residents received either the intervention or control course as part of their mandatory educational curriculum. Participating residents provided basic demographic data and information about previous communication training. They also completed the Jefferson Scale of Empathy (JSE) and Maslach Burnout Inventory (MBI), validated tools that measure empathy and burnout respectively.

Patient Participants:

Patients who had an appointment scheduled with an enrolled resident in their primary care clinic were identified through the electronic medical record (EMR). Patients with appointments scheduled at all eight clinics in our health care system were eligible to participate in the study to ensure demographic representation. Eligible patients were age 18 or older, had completed an appointment with a resident in the trial within 2 months of the resident finishing the course, and were proficient in English.

Patients were recruited by mail within two weeks of their appointment and were compensated with a $10 gift card. Survey packets contained a survey invitation cover letter, the study information sheet, the survey, and a stamped return envelope. The cover letter identified the resident the patient saw and the location of their medical appointment, to clarify which medical provider to assess in the survey. The survey consisted of the Communication Assessment Tool, the Patient Activation Measure (PAM13), and demographic questions. Three attempts were made to contact non-responders.

MEASURES

Primary Outcome - Communication Assessment Tool:

The primary outcome was a validated measure of communication, the Communication Assessment Tool (CAT). The CAT is a fifteen item survey measuring physician communication as perceived by patients. Each item is rated from 1 "Poor" to 5 "Excellent". The first fourteen items measure specific aspects of communication, and the last item measures the quality of communication overall. Because surveys such as this are subject to a ceiling effect, scores were also analyzed as the percent of questions that received the maximum score - also known as a "top box" score.

Secondary Outcomes:

In addition, the investigators evaluated whether better communication shaped patient health outcomes. Before and after the patient's clinic appointment, the investigators examined the patient's EMR and extracted information about depression, blood pressure, and admittance history. Depression was evaluated using PHQ-9 scores recorded in the EMR, a common measure of depression with well documented internal consistency and construct validity. The PHQ-9 consists of nine questions, each scored from 0 to 3 for a total score of 0 to 27, with higher scores indicating more severe depression. Scores between 5 and 10 suggest mild depression, 10-14 suggest moderate depression, and 15-27 suggest severe depression. Missed appointments ("no-shows") and cancelled appointments were recorded as the frequency per month. Hospitalizations were recorded as the frequency of hospitalization for 1, 3 and 6 months after the patient's appointment with the internal medicine resident.

Finally, patients also completed the 13-item Patient Activation Measure (PAM13), a standardized measure to assess patients' knowledge, skill, and confidence to manage their own health. Scores range from 0 (low activation) to 100 (high activation). The PAM13 was included in the patient survey.

STATISTICAL ANALYSES Summary statistics were performed for baseline characteristics both at the resident and patient levels. Frequencies with proportions were used for categorical data and means with standard deviations for continuous data. To examine the associations between intervention and control groups, the investigators used chi-square tests for categorical data, and t-tests for continuous data. At the patient level, the investigators then assessed the primary outcome, the CAT score, using multivariable logistic regression, and adjusted for gender, age, race, income, PAM-13 scores, physician's emotional exhaustion as reported on the MBI, JSE score, and year of residency. Results of models were summarized as odds ratios together with 95% Wald Confidence Intervals. All tests were 2-sided and a p<0.05 was considered statistically significant. The investigators used SAS 9.4 for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS:

* Appointment scheduled with a resident participant at one of eight primary care clinics in our health system
* had completed an appointment with a resident participant within 2 months of the resident completing their communication course
* 18 years of age or older
* proficient in English

RESIDENTS:

* PGY2 and PGY3 Internal Medicine residents at Cleveland Clinic
* Scheduled to receive required educational curriculum on communication
* Scheduled to see patients at one of the eight primary care clinics in our health system

Exclusion Criteria:

PATIENTS:

* No appointment scheduled with a resident participant at one of eight primary care clinics in our health system
* had not completed an appointment with a resident participant within 2 months of the resident completing their communication course
* Less than 18 years of age
* Not proficient in English

RESIDENTS:

* Not PGY2 and PGY3 Internal Medicine residents at Cleveland Clinic
* Not scheduled to receive required educational curriculum on communication
* Not scheduled to see patients at one of the eight primary care clinics in our health system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Communication Assessment Tool (CAT) | 2-12 weeks after primary care appointment
  The CAT is a fifteen item survey measuring physician communication as perceived by patients. Each item is rated from 1 "Poor" to 5 "Excellent". The first fourteen items measure specific aspects of communication, and the last item measures the quality of communication overall. Because surveys such as this are subject to a ceiling effect, scores were also analyzed as the percent of questions that received the maximum score - also known as a "top box" score.

SECONDARY OUTCOMES:
Patient Activation Measure (PAM13) | 2-12 weeks after primary care appointment
  PAM is a 13-item measure measure to assess patients' knowledge, skill, and confidence to manage their own health. Scores range from 0 (low activation) to 100 (high activation).

OTHER OUTCOMES:
Jefferson Scale of Empathy (JSE) | at time of resident participant recruitment
  The JSE is a 20 item 7-point Likert scale completed by the Caregiver that measures a health professional's empathy.
Maslach Burnout Inventory (MBI) | at time of resident participant recruitment
  The MBI is a 16-item survey that measures the frequency of job-related feelings of burnout using a scale of 0 (never) to 6 (every day). Burnout is measured on 3 dimensions-emotional exhaustion (EE), depersonalization (DP), and personal accomplishment (PA).

CONTACTS AND LOCATIONS:
Overall Officials: Susannah Rose, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No